CLINICAL TRIAL: NCT01176630
Title: Prevalence of Metabolic Syndrome in a Maintenance Hemodialysis Population
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Mary Schanler, Administrative Dietitian, Winthrop University Hospital
Other Study IDs: 10311
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome, ESRD patient
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is a survey to answer the specific question, "What is the prevalence of metabolic syndrome in maintenance hemodialysis patients?" Metabolic syndrome is a cluster of conditions that increase an individual's risk for developing cardiovascular disease and diabetes.

DETAILED DESCRIPTION:
Risk factors for metabolic syndrome will be collected for each consented patient. They include elevated serum triglycerides, reduced HDL cholesterol, hypertension, elevated fasting blood sugar concentration and abdominal obesity. The investigator will measure waist circumference of each consented patient in a secure area according to standardized procedures. The other data is available from the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing maintenance hemodialysis equal to or greater than 3 months
* Patient at lest 18 years of age
* Availability of all data in the medical record for classification of the metabolic syndrome, including serum triglycerides, serum HDL-cholesterol, systolic BP and diastolic BP, and serum glucose

Exclusion Criteria:

* Patients unwilling or unable to give informed consent to participate
* Patients with a history of thyroid disease
* Patients unable to stand upright

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study subjects are on maintenance hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percent of maintenance patients with at least three risk factors of metabolic syndrome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Schanler, MS, RD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital Outpatient Dialysis Unit, Mineola, New York, United States